CLINICAL TRIAL: NCT06960304
Title: Effect of a Structured Physical Exercise Program on Arteriovenous Fistula Maturation for Hemodialysis in Chronic Kidney Disease Patients
Acronym: PEFAV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unidade Local de Saúde de Coimbra, EPE (Other)
Responsible Party: Principal Investigator, CTU-CACC, Nephrology Nurse Ricardo Ferreira, Unidade Local de Saúde de Coimbra, EPE
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 035 / 24 CE
Record Dates: First submitted 2025-04-15; First posted 2025-05-07 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Disease Requiring Hemodialysis
Keywords: physical exercise; chronic kidney disease; hemodialysis; fistula maturation
MeSH Terms: conditions — Motor Activity; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercised group (Experimental): The participants in this group follow a structured physical exercise program for the arm with the Arteriovenous Fistula (AVF), including progressive exercises using weights and therapeutic balls. The goal is to assess the impact of this intervention on AVF maturation and functionality.
  Interventions: Other: Physical exercise program
- Control Group (No Intervention): The participants in this group do not follow the exercise program and only receive the usual recommendations on AVF care (standard of care).

INTERVENTIONS:
Other: Physical exercise program — Evaluation of AVF maturation using clinical and ultrasound criteria, after applying a structured physical exercise program.
  Arms: Exercised group

SUMMARY:
For patients living with Chronic Kidney Disease who are preparing to start hemodialysis, having a well-functioning arteriovenous fistula (AVF) is essential. Although the AVF is considered the best type of vascular access, its maturation process does not always go as expected-studies show that in 28% to 53% of cases, the fistula does not mature properly, making effective dialysis more difficult. There is growing interest in using physical exercise as a way to support AVF maturation. International guidelines even recommend arm exercises for this purpose. However, there is still no clear agreement on what type of exercise, how often, or how intense it should be. This study aims to evaluate whether a structured exercise program focused on the AVF arm can help improve the fistula's development and overall function.

DETAILED DESCRIPTION:
To undergo Hemodialysis (HD), it is essential for the patient to have Vascular Access (VA) for HD, with priority given to the creation of an Arteriovenous Fistula (AVF). The AVF is considered the ideal VA for HD due to its advantages over other types of access. However, to become functional, the AVF must go through a maturation process. Initial AVF maturation is a complex process of vascular adaptation and remodeling, driven by a significant increase in arterial blood flow into the vein. This requires dilation and structural changes in the blood vessel walls.

One of the main issues related to AVFs is primary maturation failure. It is estimated that between 28% and 53% of AVFs experience compromised maturation, which can hinder or even prevent effective long-term cannulation for hemodialysis treatment.

It is well recognized that physical exercise promotes vascular remodeling, as shown by increased capillarity in active muscles, the development of adjacent blood vessels, increased muscle strength, and greater diameter and prominence of veins. Due to its positive influence on vascular remodeling, exercise involving the AVF limb is frequently recommended by international best practice guidelines, and it has the potential to improve the AVF maturation process. However, current scientific evidence does not yet offer a consensus on the most effective type, duration, or intensity of exercise.

Nevertheless, intentional, repetitive, and sustained physical exercise has been shown to lead to vascular remodeling, which may positively impact the functional maturation of an AVF. In this context, the aim is to conduct a quantitative, experimental, and randomized study to evaluate the effect of implementing a Physical Exercise Program for the AVF limb (PEFAV), designed by a rehabilitation nursing specialist, on the AVF maturation process.

As part of the development of the research project titled "Effect of a Structured Physical Exercise Program on Arteriovenous Fistula Maturation", the research team intends to conduct a quantitative, experimental, and randomized study with an expected duration of twenty-four months. The main objective is to evaluate the effect of implementing a Physical Exercise Program for the AVF limb (PEFAV) on the maturation process of the AVF in individuals with stage 5 Chronic Kidney Disease (CKD) who have an upper limb AVF.

Participant recruitment will take place during the specialized nursing clinics for individuals with AV for HD at CHUC - HUC Campus, using a non-probability convenience sampling method. To ensure anonymity and data confidentiality, participants will be randomly assigned to either the Exercise Group (EG) or the Control Group (CG) through a computer-generated randomization sequence using the RedCap software, with a 1:1 allocation ratio.

Two in-person appointments with the participants will be required, both taking place at the specialized nursing clinics for CKD patients with AV for HD at CHUC - HUC Campus. During the first visit, participants will be provided with information about the study's objectives and procedures, and informed consent will be obtained. Following consent, data collection instruments and procedures will be applied. Participants in the EG will receive training and instruction on how to carry out the PEFAV, while those in the CG will receive only the usual recommendations regarding AVF care.

Each participant in the EG will receive a "PEFAV Follow-up Booklet," which will include illustrations and descriptions of the exercises, the number of sets and repetitions, and a section called the "Exercise Log," where participants will be asked to record, after each session, any sensations, perceived changes, or complications related to the AVF, as well as any difficulties performing the exercises.

At the second in-person visit (eight weeks after the first), data collection instruments and procedures will be applied again, and the EG's adherence to the PEFAV will be assessed.

Data collection will include: a questionnaire; grip strength testing and measurements of forearm and arm circumference; and data from the specialized nursing consultation report (physical examination and ultrasound criteria) at CHUC - HUC Campus.

All data collection procedures will follow formal and ethical research standards, ensuring that all informed participants voluntarily, anonymously, consent to take part in the study, with confidentiality maintained and no costs or harm to participants.

The ultimate goal is to increase the number of functional and clinically viable AVFs while reducing associated complications.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* AVF in the upper limb
* No cognitive decline and ability to follow instructions

Exclusion Criteria:

* History of previous dysfunctional ipsilateral AVF
* History of injury/condition causing pain or loss of function in the AVF limb
* Musculoskeletal conditions/osteoarticular pathology (e.g., myopathy, rheumatoid arthritis)
* Neurological conditions/cardiovascular events (e.g., stroke, peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of AVF maturation using clinical and ultrasound criteria: Diameter of the drainage vein (mm) | 8 weeks
  -Diameter of the drainage vein (mm). Eight weeks after the application of a physical exercise program, patients in the intervention and control groups will be evaluated through a physical examination (presence of thrill and continuous murmur, increased venous diameter, absence of complications such as stenosis or thrombosis) and ultrasound examination.
Evaluation of AVF maturation using clinical and ultrasound criteria: Venous wall thickness (mm) | 8 weeks
  - Venous wall thickness (mm). Eight weeks after the application of a physical exercise program, patients in the intervention and control groups will be evaluated through a physical examination (presence of thrill and continuous murmur, increased venous diameter, absence of complications such as stenosis or thrombosis) and ultrasound examination.
Evaluation of AVF maturation using clinical and ultrasound criteria: Blood velocity (cm/sec) | 8 weeks
  - Blood Velocity (cm/sec). Eight weeks after the application of a physical exercise program, patients in the intervention and control groups will be evaluated through a physical examination (presence of thrill and continuous murmur, increased venous diameter, absence of complications such as stenosis or thrombosis) and ultrasound examination.
Evaluation of AVF maturation using clinical and ultrasound criteria: Blood flow volume in the humeral artery (mL/min) | 8 weeks
  - Blood flow volume in the humeral artery (mL/min). Eight weeks after the application of a physical exercise program, patients in the intervention and control groups will be evaluated through a physical examination (presence of thrill and continuous murmur, increased venous diameter, absence of complications such as stenosis or thrombosis) and ultrasound examination.

SECONDARY OUTCOMES:
Evaluation of the impact of each physical parameters in FAV maturation: Change in Handgrip Strength (kg) | 8 weeks
  The Change in Handgrip Strength will be measured: kg
Evaluation of the impact of each physical parameters in FAV maturation: Change in Forearm and Upper Arm Circumference (cm) | 8 weeks
  The Change in Forearm and Upper Arm Circumference will be measured: cm
Evaluation of the impact of each physical parameters in FAV maturation: Change in Rate of AVF Complications (%) | 8 weeks
  The Change in Rate of AVF Complications will be measured: %
Evaluation of the impact of each physical parameters in FAV maturation: Change in Blood Flow Velocity in the Humeral Artery (mL/min) | 8 weeks
  The change in Blood Flow Velocity in the Humeral Artery will be measured: mL/min.
Evaluation of adherence Rate to the Exercise Program for the AVF Limb (%) | Within 7 weeks
  The percentage of exercise group participants who consistently completed the program will be assessed, based on daily records and weekly phone contacts. Participants will be further classified according to different adherence levels to the physical program (low, moderate, and high), based on the number of entries in the tracking diary.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo A. S. Ferreira, Bachelor's degree in Nursing, Principal Investigator — Unidade Local de Saude de Coimbra
Locations (1):
- Unidade Local de Saude de Coimbra, Coimbra, Coimbra District, Portugal

IPD SHARING:
Plan to Share IPD: No
Data will be irreversibly anonymized and exclusively handled by researchers involved in the study.